CLINICAL TRIAL: NCT01250496
Title: A Randomized Double-Blind Placebo Controlled Study With Aminophylline to Attenuate the Side Effect Profile of Regadenoson in Patients Undergoing Myocardial Perfusion Imaging.
Brief Title: Study With Aminophylline to Attenuate of the Side Effects of Regadenoson
Acronym: ASSUAGE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to nationwide shortage of Aminophylline. Enrolled subjects did not complete study.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Rami Doukky, Director of Nuclear Cardiology and Stress Testing Laboratories, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASSUAGETrial
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Patients Being Assessed With Nuclear Stress Testing of the Heart Using the Stress Agent Regadenoson, Lexiscan
Keywords: regadenoson; lexiscan; aminophylline; SPECT; Myocardial Perfusion Imaging; pharmacologic stress test
MeSH Terms: interventions — Aminophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline (Experimental): 75 mg of intravenous aminophylline.
  Interventions: Drug: Aminophylline
- Placebo (Placebo Comparator): Matching normal saline placebo (sterile salt water).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminophylline — 75 mg of intravenous aminophylline
  Arms: Aminophylline
Drug: Placebo — Matching 0.9 Normal Saline (sterile salt water)administered intravenously.
  Arms: Placebo

SUMMARY:
The routine administration of 75 mg of intravenous aminophylline following regadenoson (Lexiscan®), a commonly used medication for nuclear stress testing of the heart, can reduce the gastrointestinal (diarrhea and stomach upset) and other side effects related to regadenoson.

DETAILED DESCRIPTION:
Approximately 250 patients who are referred for a nuclear stress testing of the heart with regadenoson (Lexiscan®) will be recruited to participate in the study. Following regadenoson (administered as part of a stress routine test protocol) participants will receive either aminophylline (75 mg - intravenously) or a matching inactive placebo (sterile salt water) injection. Participants will be surveyed for gastrointestinal symptoms and other side effects related to regadenoson. The frequency and severity of such side effects will be compared between the two study groups (aminophylline vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred to undergo a clinically-indicated regadenoson-stress myocardial perfusion imaging at Rush University Medical Center

Exclusion Criteria:

* Patient refusal to participate
* Known allergic reaction to aminophylline.
* Pre-existing headache or acute/subacute GI illness with symptoms of diarrhea, abdominal discomfort, nausea or vomiting.
* Any contraindication to aminophylline: hypotension, unstable cardiac arrhythmias and acute coronary symptoms.
* Uncontrolled seizure disorder defined as more than 2 seizure episodes in the past 12 months or any seizure in the past week.
* Pregnant or breast-feeding women.
* Patients receiving anti-platelet agent dipyridamole (Persantine® or Aggrenox®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Doukky R, Morales Demori R, Jain S, Kiriakos R, Mwansa V, Calvin JE. Attenuation of the side effect profile of regadenoson: a randomized double-blinded placebo-controlled study with aminophylline in patients undergoing myocardial perfusion imaging. "The ASSUAGE trial". J Nucl Cardiol. 2012 Jun;19(3):448-57. doi: 10.1007/s12350-012-9533-x. Epub 2012 Mar 7. PMID 22395779
- [Derived] Ballany W, Mansour K, Morales Demori R, Al-Amoodi M, Doukky R. The impact of regimented aminophylline use on extracardiac radioisotope activity in patients undergoing regadenoson stress SPECT myocardial perfusion imaging: a substudy of the ASSUAGE trial. J Nucl Cardiol. 2014 Jun;21(3):496-502. doi: 10.1007/s12350-014-9864-x. Epub 2014 Feb 12. PMID 24519563
- See also: Pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/22395779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the stress testing laboratories of Rush University Medical Center in the period from November 23, 2010 through February 10, 2011.
Pre-assignment Details: Two consenting subjects did not undergo regadenoson-stress for a clinical reason and were subsequently excluded.
  Otherwise, the remainder of connecting patients received the intervention they are allocated to, completed follow-up and analyzed within the group they were randomized to.
Period: Overall Study
Arm/Group | Aminophylline | Placebo
Started | 124 | 124
Completed | 0 | 0
Not Completed | 124 | 124
Not completed — Study terminated | 124 | 124

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aminophylline | Placebo | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 56 | 109
  >=65 years | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.1) | 62.0 (13.6) | 62.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 54 | 111
  Male | 67 | 70 | 137
Region of Enrollment [Number; unit: participants]
  United States | 124 | 124 | 248

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoints of Abdominal Cramps and Diarrhea.
Description: Patients will be surveyed for these symptoms following to the completion of the cardiac stress testing procedure and prior to discharge from the laboratory.
Time Frame: within 2 hours from the intervention.
Population: All enrolled patients who received the intervention (n=248; 124 aminophylline ans 124 placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 124 | 124
Participants | 11 | 22
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; null hypothesis: aminophylline administration does not reduce the incidence of the primary endpoint as compared to placebo. The chi-square test was used to compare event rate between the study arm; Test type: Superiority or Other; p = 0.04, Chi-squared — No adjustment for multiple comparisons was performed. The threshold for statistical significance was < 0.05; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.2 to 0.98]

2. Secondary Outcome: "Number of Participants With Composite Endpoint of Any Regadenoson-related Side Effects.
Description: The secondary end-point encompasses any one (or more) regadenoson-related side effects of flushing /feeling hot, chest pain /chest discomfort, angina, headache, dizziness, abdominal cramps/discomfort, diarrhea, and/or nausea.
  If multiple side effects occur only one side effect is counted.
Time Frame: within 2 hours from the intervention.
Population: All enrolled patients who received the intervention (n= 248; 124 aminophyllineand and 124 placebo).
Measure: Number; unit: participants
Arm/Group | Aminophylline | Placebo
Number analyzed (Participants) | 124 | 124
participants | 55 | 83
Statistical Analysis 1: Comparison: Aminophylline vs Placebo; null hypothesis: the rate of regadenoson adverse effects (global symptomatic burden) in the aminophylline and placebo group are not statistically different. The chi-square test was used for comparison; Test type: Superiority or Other; p < 0.001, Chi-squared — P value is not adjusted for multiple comparisons; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.2 to 0.7]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Clinically determined adverse events that require treatment
Arm/Group | Aminophylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/124
Other Adverse Events (participants affected / at risk) | 55/124 | 83/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminophylline (N=124) | Placebo (N=124)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) — Any treatment-requiring tachyarrhythmia that was not present at baseline occurring in the 24 hours ensuing the regadenoson stress test.
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) — Events of cardiac arrest due to ventricular tachycardia, ventricular fibrillation, asystole, or pulseless electrical activity that lead to the initiation of Advanced Cardiac Life Support protocol in the 24 hours ensuing the regadenoson stress test.
Hospitalization (General disorders) | 0 (0) | 0 (0) — Any event leading to patient hospitalization from any cause in the 24 hours ensuing the regadenoson stress test.
Seizure (Nervous system disorders) | 0 (0) | 0 (0) — Any seizure event in the 24 hours ensuing the regadenoson stress test.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Bronchospasm or auscultatory wheezing with shortness of breath occurring in the 24 hours following regadenoson administration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aminophylline (N=124) | Placebo (N=124)
Flushing (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6) — Flushing sensation occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 23 (23) — Dyspnea sensation occuring any time after the administration of regadenoson until the patient's dismissal from the nuclear laboratory.
Headache (Nervous system disorders) | 9 (9) | 31 (31) — Headache symptoms occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Chest discomfort or pain (Cardiac disorders) | 13 (13) | 15 (15) — Chest discomfort occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Angina (Cardiac disorders) | 0 (0) | 0 (0) — Angina symptoms occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Feeling hot (Skin and subcutaneous tissue disorders) | 11 (11) | 12 (12) — Hot sensation occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Nausea (Gastrointestinal disorders) | 21 (21) | 22 (22) — Nausea occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Abdominal cramp or discomfort (Gastrointestinal disorders) | 10 (10) | 17 (17) — Abdominal cramps or discomfort occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Dizziness (Nervous system disorders) | 31 (31) | 45 (45) — Dizziness symptoms occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Diarrhea (Gastrointestinal disorders) | 4 (4) | 13 (13) — Diarrhea or loose bowel movement occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Open label aminophylline use (Injury, poisoning and procedural complications) | 1 (1) | 7 (7) — Intravenous aminophylline to treat regadenoson-related side effects, administered after regadenoson injection
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) — Self-limiting atrial fibrillation, not requiring treatment, occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) — Self-limiting supraventricular tachycardia, not requiring treatment, occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) — Self-limiting non-sustained ventricular tachycardia, not requiring treatment, occurring anytime after the administration of regadenoson until the patient's dismissal from the nuclear laboratory

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No